CLINICAL TRIAL: NCT03245008
Title: A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients With Osteoarthritis Accompanied by Moderate to Severe Pain
Brief Title: Efficacy and Safety of MT-5547 in Patients With Osteoarthritis Accompanied by Moderate to Severe Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-5547-J01
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee / Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MT-5547 dosing regimen 1 (Experimental): MT-5547 Subcutaneous (SC) dosing regimen 1. Naproxen-matching placebo oral after Week 16.
  Interventions: Drug: MT-5547
- MT-5547 dosing regimen 2 (Experimental): MT-5547 SC dosing regimen 2. Naproxen-matching placebo oral after Week 16.
  Interventions: Drug: MT-5547; Drug: MT-5547-matching placebo
- MT-5547-matching placebo (Placebo Comparator): MT-5547-matching placebo SC dosing. Naproxen oral after Week 16.
  Interventions: Drug: MT-5547-matching placebo

INTERVENTIONS:
Drug: MT-5547 — Solution for injection in pre-filled syringe
  Other Names: Fasinumab
  Arms: MT-5547 dosing regimen 1; MT-5547 dosing regimen 2
Drug: MT-5547-matching placebo — Solution for injection in pre-filled syringe
  Arms: MT-5547 dosing regimen 2; MT-5547-matching placebo

SUMMARY:
The objective of this study is to verify the superiority of 16 weeks of MT-5547 treatment to placebo, as evidenced by the WOMAC pain score (the efficacy outcome measure), in patients with osteoarthritis of the knee or hip. Additional objectives of the study are to investigate the efficacy, safety, and pharmacokinetics of MT-5547 in long-term use.

DETAILED DESCRIPTION:
The blind will be maintained, including for the study sponsor, until the key code is opened after the data have been fixed for all subjects in Week 24. In addition, in order to eliminate any bias that could affect the study assessments, to the extent possible, the blind will be maintained with respect to the study site and the subject even after the opening of the study sponsor key code.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Male and female Japanese patients, 40 years to 85 years at the time written informed consent is obtained.
* Patients who have been diagnosed with osteoarthritis (OA) of the knee or hip based on the American College of Rheumatology (ACR) criteria.
* Patients with an evaluated joint (knee or hip) with a K-L (Kellgren-Lawrence) score of ≥2 based on the X-ray test performed.
* Moderate to severe pain in the evaluated joint, defined as a WOMAC pain score of ≥4 (mean of the 5 items), on the WOMAC assessments.
* Patients who satisfy both 1) and 2) below.

  1. Inadequate OA pain relief from at least 1 oral NSAID.
  2. Intolerance to or inadequate OA pain relief from at least 1 opioid (including combination drugs), or unwillingness to take opioid therapy.
* Patients who agree to not change their current lifestyle (daily living activities and exercise) throughout the study.
* Patients who are able to complete post-operative follow-up for any joint replacement surgery that is performed during the study.
* Body mass index at screening ≤39.
* Patient who are able to understand and answer endpoint questions used in the study.

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Presence of symptoms of carpal tunnel syndrome within 6 months before screening.
* Patients who cannot undergo MRI.
* Trauma to the index joint within 3 months prior to screening.
* Presence or history of inflammatory joint diseases other than OA, Paget's disease of the spine, pelvis or femur, multiple sclerosis, fibromyalgia, vertebral tumors or infections, or renal osteodystrophy.
* Presence or history, confirmed by imaging, of arthropathy, neuropathic joint arthropathy, hip dislocation, knee dislocation, extensive subchondral cyst, marked bone destruction or bone loss, or pathologic fractures.
* Autonomic neuropathy diagnosed in the assessment of autonomic nerve symptoms performed at screening, or baseline.
* Presence or history of orthostatic hypotension at the orthostatic hypotension assessments performed at screening, prerandomization, or baseline.
* Presence or history of autonomic neuropathy, diabetic neuropathy, or other peripheral neuropathy such as reflex sympathetic dystrophy at screening.
* Presence or history of chronic familial dysautonomia.
* Intolerance to naproxen.
* Systemic (excluding topical, intranasal, ophthalmic, and inhaled formulations) corticosteroids within 4 weeks prior to screening.
* Intra-articular corticosteroids in the evaluated joint within 12 weeks prior to screening, or in any other joint within 4 weeks prior to screening.
* Received an intra-articular injection of hyaluronic acid in any joint within the period specified for each medicine prior to screening.
* Resting heart rate of <50 bpm or >100 bpm at screening, or baseline.
* Presence or history of 2nd or 3rd degree heart block, 1st degree heart block with abnormal QRS, or bifascicular block by ECG assessment at screening.
* Non-compliance with the Numerical rating scale (NRS) recording (average pain on walking in the evaluated joint over 1 day) during the pre-treatment observation period.
* Women who are pregnant, breast-feeding, or may be pregnant.
* Use of an anti-Nerve growth factor (anti-NGF) antibody in the past, or apparent hypersensitivity or intolerance to anti-NGF antibodies.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (27):
- Japan (27):
  - Investigational Site, Aichi
  - Investigational Site, Aomori
  - Investigational Site, Chiba
  - Investigational Site, Ehime
  - Investigational Site, Fukui
  - Investigational Site, Fukuoka
  - Investigational Site, Fukushima
  - Investigational Site, Gunma
  - Investigational Site, Hiroshima
  - Investigational Site, Hokkaido
  - Investigational Site, Hyōgo
  - Investigational Site, Ibaraki
  - Investigational Site, Kagoshima
  - Investigational Site, Kanagawa
  - Investigational Site, Kumamoto
  - Investigational Site, Kyoto
  - Investigational Site, Mie
  - Investigational Site, Miyagi
  - Investigational Site, Miyazaki
  - Investigational Site, Osaka
  - Investigational Site, Ōita
  - Investigational Site, Saitama
  - Investigational Site, Shiga
  - Investigational Site, Shizuoka
  - Investigational Site, Tokyo
  - Investigational Site, Yamagata
  - Investigational Site, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Groups:
- Pooled Placebo: This group consists of total of 204 participants who were randomized to Placebo group before (N=39) and after (N=165) the protocol amendment.
  Participants randomized to this group received MT-5547-matching placebo SC q4w from Week 0 to Week 44.
  Naproxen oral was received from the day after the Week 16 until Week 48.
- Pooled MT-5547 1 mg q4w: This group consists of total 203 participants who were randomized to MT-5547 1 mg q4w group before (N=38) and after (N=165) the protocol amendment.
  Participants randomized to this group received MT-5547 1 mg SC q4w from Week 0 to Week 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- After the Amendment MT-5547 1 mg q8w: This group was added after Protocol Amendment. Participants randomized to this group received MT-5547 1 mg SC on Weeks 0, 8, 16, 24, 32, and 40, and MT-5547-matching placebo SC on Weeks 4, 12, 20, 28, 36, and 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 3 mg q4w: This group was removed from this study dosing regimen after protocol amendment. Participants randomized to the MT-5547 3 mg q4w group received MT-5547 3 mg SC q4w from Week 0 to Week 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 6 mg q8w: This group was removed from this study dosing regimen after protocol amendment. Participants randomized to the After the amendment MT-5547 6 mg q8w group received MT-5547 6 mg SC on Weeks 0, 8, 16, 24, 32, and 40, and MT-5547-matching placebo SC on Weeks 4, 12, 20, 28, 36, and 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
Period: Overall Study
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment MT-5547 1 mg q8w | MT-5547 3 mg q4w | MT-5547 6 mg q8w
Started | 204 | 203 | 162 | 28 | 29
Completed | 164 | 159 | 132 | 0 | 0
Not Completed | 40 | 44 | 30 | 28 | 29
Not completed — Adverse Event | 15 | 18 | 15 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 3 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 19 | 11 | 0 | 0
Not completed — Discontinuation of 3 mg q4w and 6 mg q8w doses | 0 | 0 | 0 | 27 | 27
Not completed — Failure to meet randomization criteria | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The pooled placebo group (N=204) and the pooled MT-5547 1 mg q4w group (N=203) showed the total number of participants randomized to each group before and after the protocol amendment.
  The number of participants who were randomized to the placebo group (N=165) and the MT-5547 1 mg q4w group (N=165) after the protocol amendment were not shown in the table below because they are included in the respective pooled groups. A total of 626 participants were enrolled into this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment MT-5547 1 mg q8w | MT-5547 3 mg q4w | MT-5547 6 mg q8w | Total
Number analyzed (Participants) | 204 | 203 | 162 | 28 | 29 | 626
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.4) | 66.1 (9.7) | 66.6 (9.4) | 68.6 (7.6) | 65.2 (7.4) | 66.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 160 | 126 | 20 | 25 | 494
  Male | 41 | 43 | 36 | 8 | 4 | 132
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 204 | 203 | 162 | 28 | 29 | 626
BMI [Mean (Standard Deviation); unit: kg/㎡] | 26.6 (4.3) | 27.0 (4.4) | 26.8 (4.2) | 24.8 (3.4) | 27.3 (4.5) | 26.8 (4.3)
Index Joint [Count of Participants; unit: Participants] — The index joint was the joint (knee or hip) that was judged to have a K-L score of ≥2 in the X-ray (centralized assessment) and the joint with the highest WOMAC pain subscale score (mean of 5 items).
  Participants
    Knee | 189 | 190 | 150 | 26 | 26 | 581
    Hip | 15 | 13 | 12 | 2 | 3 | 45
K-L Score [Count of Participants; unit: Participants] — Kellgren-Lawrence category. Osteoarthritis staging category based on simple X-ray; a 5-level scale from 0 to 4. Higher scores indicated worse.
  Participants
    1 | 0 | 0 | 0 | 0 | 0 | 0
    2 | 39 | 36 | 24 | 2 | 3 | 104
    3 | 95 | 97 | 82 | 15 | 15 | 304
    4 | 70 | 70 | 56 | 11 | 11 | 218
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The WOMAC is a scale that is used to assess the activities of daily living in osteoarthritis, the WOMAC pain subscale score was defined as the average of 5 items (during walking, using stairs, in bed, sitting or lying, and standing). The participants assessed the past 48 hours on an 11-point numeric rating scale, from 0 (no pain) to 10 (worst pain imaginable), where higher scores indicated worse pain.
  units on a scale | 5.93 (1.33) | 6.01 (1.31) | 6.02 (1.39) | 6.32 (1.51) | 6.34 (1.29) | 6.02 (1.35)

OUTCOME MEASURES:

1. Primary Outcome: WOMAC Pain Score (Change From Baseline at Week 16)
Description: The WOMAC is a scale that is used to assess the activities of daily living in osteoarthritis, the WOMAC pain subscale score was defined as the average of 5 items (during walking, using stairs, in bed, sitting or lying, and standing). The participants assessed the past 48 hours on an 11-point numeric rating scale, from 0 (no pain) to 10 (worst pain imaginable), where higher scores indicated worse pain.
Time Frame: Baseline to Week 16
Population: Analysis was performed on modified FAS(mFAS). For the analysis of After amendment MT-5547 1 mg ｑ8w group comparing to placebo group and MT-5547 1 mg q4w group, after the protocol amendment randomized populations are also presented. This study produced 16-week treatment period dataset, 24-week treatment period dataset, and 68-week treatment period dataset. The results in this section are presented in the 16-week treatment period dataset.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- After the Amendment Placebo: Participants in this group were randomized to Placebo group after the protocol amendment. Participants randomized to this group received MT-5547-matching placebo SC q4w from Week 0 to Week 44.
  Naproxen oral was received from the day after the Week 16 until Week 48. These participants were included in the Pooled Placebo group.
- After the Amendment MT-5547 1 mg q4w: Participants in this group were randomized to MT-5547 1mg q4w group after the protocol amendment.
  Participants randomized to this group received MT-5547 1 mg SC q4w from Week 0 to Week 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
  These participants were included in the pooled MT-5547 1mg q4w group.
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment Placebo | After the Amendment MT-5547 1 mg q8w | After the Amendment MT-5547 1 mg q4w
Number analyzed (Participants) | 204 | 203 | 165 | 162 | 165
units on a scale | -1.74 (0.17) | -2.96 (0.17) | -1.78 (0.18) | -2.12 (0.18) | -2.79 (0.18)
Statistical Analysis 1: Comparison: Pooled Placebo vs Pooled MT-5547 1 mg q4w; Test type: Superiority; p < 0.001, Mixed Models Analysis — Adjusted P-value; Least Squares Mean Difference = -1.22, 95% CI 2-sided [-1.57 to -0.86], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: After the Amendment Placebo vs After the Amendment MT-5547 1 mg q8w; Test type: Superiority; p = 0.103, Mixed Models Analysis — Adjusted P-value; Least Squares Mean Difference = -0.34, 95% CI 2-sided [-0.76 to 0.07], Standard Error of Mean 0.21

2. Secondary Outcome: WOMAC Physical Function Score (Change From Baseline at Week 16)
Description: The WOMAC physical function subscale score was defined as the average of 17 items(the level of difficulty of activities of daily living: stair use, rising from sitting, standing, bending, walking, getting in and out of a car, shopping, putting on and taking off socks, rising from bed, lying in bed, getting in and out of the bath, sitting, getting on and off the toilet, heavy household duties, light household duties). The participants assessed the past 48 hours on an 11-point numeric rating scale, from 0 (no difficulty) to 10(extremely difficult), where higher scores indicated worse function limitation.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment Placebo | After the Amendment MT-5547 1 mg q8w | After the Amendment MT-5547 1 mg q4w
Number analyzed (Participants) | 204 | 203 | 165 | 162 | 165
units on a scale | -1.38 (0.16) | -2.64 (0.16) | -1.44 (0.17) | -1.88 (0.17) | -2.53 (0.17)
Statistical Analysis 1: Comparison: Pooled Placebo vs Pooled MT-5547 1 mg q4w; Test type: Superiority; p < 0.001, Mixed Models Analysis — Adjusted P-value; Least Squares Mean Difference = -1.26, 95% CI 2-sided [-1.60 to -0.92], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: After the Amendment Placebo vs After the Amendment MT-5547 1 mg q8w; Test type: Superiority; Least Squares Mean Difference = -0.45, 95% CI 2-sided [-0.84 to -0.05], Standard Error of Mean 0.20

3. Secondary Outcome: WOMAC Pain Score (Change From Baseline at Each Assessment Time Point)
Description: as for outcome 1
Time Frame: Baseline to Week 68
Population: Analysis was performed on modified FAS(mFAS). For the analysis of After amendment MT-5547 1 mg ｑ8w group comparing to placebo group and MT-5547 1 mg q4w group, after the protocol amendment randomized populations are also presented. This study produced 16-week, 24-week, and 68-week treatment period datasets. The results in this section are presented in the 68-week treatment period dataset. Here 'n' = Number of evaluable participants at the specified point in time.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment Placebo | After the Amendment MT-5547 1 mg q8w | After the Amendment MT-5547 1 mg q4w
Number analyzed (Participants) | 204 | 203 | 165 | 162 | 165
units on a scale
  Week 1: number analyzed (Participants) | 203 | 203 | 165 | 162 | 165
  Week 1 | -0.63 (0.14) | -1.52 (0.14) | -0.58 (0.14) | -1.22 (0.15) | -1.40 (0.14)
  Week 2: number analyzed (Participants) | 201 | 200 | 162 | 162 | 162
  Week 2 | -0.80 (0.15) | -1.80 (0.15) | -0.78 (0.15) | -1.55 (0.15) | -1.65 (0.15)
  Week 4: number analyzed (Participants) | 201 | 201 | 163 | 162 | 163
  Week 4 | -1.03 (0.15) | -2.10 (0.16) | -0.98 (0.16) | -1.68 (0.16) | -1.90 (0.16)
  Week 8: number analyzed (Participants) | 199 | 200 | 161 | 160 | 162
  Week 8 | -1.29 (0.16) | -2.65 (0.16) | -1.26 (0.17) | -1.76 (0.17) | -2.45 (0.17)
  Week 12: number analyzed (Participants) | 193 | 197 | 155 | 158 | 159
  Week 12 | -1.62 (0.17) | -2.77 (0.17) | -1.61 (0.18) | -2.27 (0.18) | -2.56 (0.18)
  Week 16: number analyzed (Participants) | 190 | 189 | 152 | 158 | 152
  Week 16 | -1.75 (0.17) | -2.97 (0.17) | -1.76 (0.18) | -2.10 (0.18) | -2.77 (0.18)
  Week 20: number analyzed (Participants) | 189 | 185 | 151 | 157 | 150
  Week 20 | -2.43 (0.17) | -3.06 (0.17) | -2.38 (0.18) | -2.54 (0.18) | -2.85 (0.18)
  Week 24: number analyzed (Participants) | 186 | 180 | 148 | 149 | 146
  Week 24 | -2.54 (0.18) | -3.04 (0.18) | -2.52 (0.18) | -2.39 (0.18) | -2.90 (0.19)
  Week 28: number analyzed (Participants) | 184 | 177 | 146 | 143 | 143
  Week 28 | -2.50 (0.18) | -3.19 (0.18) | -2.48 (0.18) | -2.83 (0.18) | -3.05 (0.18)
  Week 32: number analyzed (Participants) | 180 | 175 | 142 | 142 | 141
  Week 32 | -2.62 (0.18) | -3.29 (0.18) | -2.63 (0.18) | -2.60 (0.18) | -3.13 (0.18)
  Week 36: number analyzed (Participants) | 173 | 173 | 135 | 136 | 139
  Week 36 | -2.66 (0.18) | -3.16 (0.18) | -2.72 (0.18) | -2.84 (0.18) | -2.99 (0.18)
  Week 40: number analyzed (Participants) | 170 | 171 | 133 | 133 | 137
  Week 40 | -2.68 (0.18) | -3.28 (0.18) | -2.70 (0.19) | -2.74 (0.19) | -3.08 (0.19)
  Week 44: number analyzed (Participants) | 170 | 162 | 133 | 134 | 129
  Week 44 | -2.72 (0.18) | -3.25 (0.18) | -2.74 (0.18) | -3.03 (0.18) | -3.03 (0.19)
  Week 48: number analyzed (Participants) | 170 | 161 | 133 | 132 | 128
  Week 48 | -2.75 (0.19) | -3.17 (0.19) | -2.75 (0.19) | -2.77 (0.19) | -2.99 (0.19)
  Week 52: number analyzed (Participants) | 167 | 160 | 131 | 133 | 127
  Week 52 | -2.35 (0.19) | -2.80 (0.20) | -2.43 (0.20) | -2.42 (0.20) | -2.56 (0.20)
  Week 60: number analyzed (Participants) | 163 | 156 | 127 | 131 | 123
  Week 60 | -2.53 (0.20) | -2.02 (0.20) | -2.61 (0.21) | -2.32 (0.21) | -1.78 (0.21)
  Week 68: number analyzed (Participants) | 162 | 151 | 126 | 130 | 121
  Week 68 | -2.49 (0.20) | -2.05 (0.21) | -2.60 (0.20) | -2.38 (0.20) | -1.84 (0.21)

4. Secondary Outcome: WOMAC Physical Function Score (Change From Baseline at Each Assessment Time Point)
Description: as for outcome 2
Time Frame: Baseline to Week 68
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment Placebo | After the Amendment MT-5547 1 mg q8w | After the Amendment MT-5547 1 mg q4w
Number analyzed (Participants) | 204 | 203 | 165 | 162 | 165
units on a scale
  Week 1: number analyzed (Participants) | 203 | 203 | 165 | 162 | 165
  Week 1 | -0.44 (0.14) | -1.23 (0.14) | -0.4 (0.14) | -0.98 (0.14) | -1.12 (0.14)
  Week 2: number analyzed (Participants) | 201 | 200 | 162 | 162 | 162
  Week 2 | -0.56 (0.14) | -1.55 (0.14) | -0.52 (0.14) | -1.25 (0.14) | -1.41 (0.14)
  Week 4: number analyzed (Participants) | 201 | 201 | 163 | 162 | 163
  Week 4 | -0.73 (0.15) | -1.81 (0.15) | -0.71 (0.15) | -1.38 (0.15) | -1.64 (0.15)
  Week 8: number analyzed (Participants) | 199 | 200 | 161 | 160 | 162
  Week 8 | -0.97 (0.15) | -2.34 (0.16) | -0.94 (0.16) | -1.48 (0.16) | -2.17 (0.16)
  Week 12: number analyzed (Participants) | 193 | 197 | 155 | 158 | 159
  Week 12 | -1.26 (0.16) | -2.43 (0.16) | -1.22 (0.17) | -1.94 (0.17) | -2.23 (0.17)
  Week 16: number analyzed (Participants) | 190 | 189 | 152 | 158 | 152
  Week 16 | -1.40 (0.16) | -2.66 (0.16) | -1.40 (0.17) | -1.84 (0.17) | -2.49 (0.17)
  Week 20: number analyzed (Participants) | 189 | 185 | 151 | 157 | 150
  Week 20 | -2.02 (0.16) | -2.74 (0.16) | -1.95 (0.17) | -2.20 (0.17) | -2.53 (0.17)
  Week 24: number analyzed (Participants) | 186 | 180 | 148 | 149 | 146
  Week 24 | -2.22 (0.17) | -2.74 (0.17) | -2.17 (0.18) | -2.02 (0.18) | -2.61 (0.18)
  Week 28: number analyzed (Participants) | 184 | 177 | 146 | 143 | 143
  Week 28 | -2.18 (0.17) | -2.90 (0.17) | -2.15 (0.17) | -2.41 (0.17) | -2.76 (0.17)
  Week 32: number analyzed (Participants) | 180 | 175 | 142 | 142 | 141
  Week 32 | -2.22 (0.17) | -3.00 (0.17) | -2.23 (0.17) | -2.23 (0.17) | -2.83 (0.17)
  Week 36: number analyzed (Participants) | 173 | 173 | 135 | 136 | 139
  Week 36 | -2.31 (0.17) | -2.84 (0.17) | -2.33 (0.17) | -2.47 (0.17) | -2.67 (0.17)
  Week 40: number analyzed (Participants) | 170 | 171 | 133 | 133 | 137
  Week 40 | -2.29 (0.17) | -2.91 (0.17) | -2.29 (0.18) | -2.46 (0.18) | -2.71 (0.18)
  Week 44: number analyzed (Participants) | 170 | 162 | 133 | 134 | 129
  Week 44 | -2.35 (0.17) | -2.90 (0.17) | -2.37 (0.17) | -2.67 (0.18) | -2.69 (0.18)
  Week 48: number analyzed (Participants) | 170 | 161 | 133 | 132 | 128
  Week 48 | -2.38 (0.18) | -2.83 (0.18) | -2.35 (0.18) | -2.46 (0.18) | -2.61 (0.18)
  Week 52: number analyzed (Participants) | 167 | 160 | 131 | 133 | 127
  Week 52 | -2.03 (0.18) | -2.51 (0.19) | -2.06 (0.19) | -2.10 (0.19) | -2.26 (0.19)
  Week 60: number analyzed (Participants) | 163 | 156 | 127 | 131 | 123
  Week 60 | -2.18 (0.19) | -1.75 (0.19) | -2.22 (0.20) | -1.98 (0.20) | -1.52 (0.20)
  Week 68: number analyzed (Participants) | 162 | 151 | 126 | 130 | 121
  Week 68 | -2.14 (0.19) | -1.71 (0.20) | -2.22 (0.20) | -2.10 (0.20) | -1.51 (0.20)

5. Secondary Outcome: WOMAC Stiffness Score (Change From Baseline at Each Assessment Time Point)
Description: The WOMAC stiffness subscale score was defined as the average of 2 items(after first waking and later in the day). The participants assessed the past 48 hours on an 11-point numeric rating scale, from 0 (no stiffness) to 10(extremely stiffness), where higher scores indicated worse stiffness.
Time Frame: Baseline to Week 68
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment Placebo | After the Amendment MT-5547 1 mg q8w | After the Amendment MT-5547 1 mg q4w
Number analyzed (Participants) | 204 | 203 | 165 | 162 | 165
units on a scale
  Week 1: number analyzed (Participants) | 203 | 203 | 165 | 162 | 165
  Week 1 | -0.24 (0.15) | -1.21 (0.15) | -0.24 (0.15) | -0.97 (0.15) | -1.21 (0.15)
  Week 2: number analyzed (Participants) | 201 | 200 | 162 | 162 | 162
  Week 2 | -0.42 (0.16) | -1.55 (0.16) | -0.45 (0.16) | -1.26 (0.16) | -1.56 (0.16)
  Week 4: number analyzed (Participants) | 201 | 201 | 163 | 162 | 163
  Week 4 | -0.58 (0.16) | -1.78 (0.16) | -0.62 (0.17) | -1.37 (0.17) | -1.73 (0.17)
  Week 8: number analyzed (Participants) | 199 | 200 | 161 | 160 | 162
  Week 8 | -0.72 (0.17) | -2.29 (0.17) | -0.75 (0.17) | -1.47 (0.18) | -2.24 (0.18)
  Week 12: number analyzed (Participants) | 193 | 197 | 155 | 158 | 159
  Week 12 | -0.99 (0.17) | -2.36 (0.18) | -1.01 (0.18) | -1.94 (0.18) | -2.30 (0.18)
  Week 16: number analyzed (Participants) | 190 | 189 | 152 | 158 | 152
  Week 16 | -1.21 (0.17) | -2.63 (0.18) | -1.24 (0.18) | -1.78 (0.18) | -2.58 (0.18)
  Week 20: number analyzed (Participants) | 189 | 185 | 151 | 157 | 150
  Week 20 | -1.93 (0.17) | -2.74 (0.18) | -1.95 (0.18) | -2.21 (0.18) | -2.65 (0.18)
  Week 24: number analyzed (Participants) | 186 | 180 | 148 | 149 | 146
  Week 24 | -2.13 (0.17) | -2.80 (0.18) | -2.16 (0.18) | -1.86 (0.18) | -2.74 (0.19)
  Week 28: number analyzed (Participants) | 184 | 177 | 146 | 143 | 143
  Week 28 | -2.02 (0.17) | -2.96 (0.18) | -2.01 (0.18) | -2.31 (0.18) | -2.89 (0.18)
  Week 32: number analyzed (Participants) | 180 | 175 | 142 | 142 | 141
  Week 32 | -2.22 (0.18) | -2.94 (0.18) | -2.31 (0.19) | -2.19 (0.19) | -2.86 (0.19)
  Week 36: number analyzed (Participants) | 173 | 173 | 135 | 136 | 139
  Week 36 | -2.16 (0.18) | -2.91 (0.18) | -2.23 (0.18) | -2.53 (0.18) | -2.87 (0.18)
  Week 40: number analyzed (Participants) | 170 | 171 | 133 | 133 | 137
  Week 40 | -2.16 (0.18) | -2.97 (0.18) | -2.24 (0.18) | -2.44 (0.18) | -2.92 (0.18)
  Week 44: number analyzed (Participants) | 170 | 162 | 133 | 134 | 129
  Week 44 | -2.29 (0.18) | -3.01 (0.18) | -2.38 (0.18) | -2.56 (0.18) | -2.93 (0.18)
  Week 48: number analyzed (Participants) | 170 | 161 | 133 | 132 | 128
  Week 48 | -2.27 (0.19) | -2.87 (0.19) | -2.34 (0.19) | -2.34 (0.19) | -2.81 (0.19)
  Week 52: number analyzed (Participants) | 167 | 160 | 131 | 133 | 127
  Week 52 | -1.83 (0.20) | -2.51 (0.20) | -1.93 (0.20) | -1.98 (0.20) | -2.44 (0.20)
  Week 60: number analyzed (Participants) | 163 | 156 | 127 | 131 | 123
  Week 60 | -2.06 (0.21) | -1.51 (0.21) | -2.17 (0.21) | -1.85 (0.21) | -1.45 (0.21)
  Week 68: number analyzed (Participants) | 162 | 151 | 126 | 130 | 121
  Week 68 | -2.09 (0.21) | -1.49 (0.21) | -2.23 (0.21) | -1.90 (0.21) | -1.44 (0.22)

6. Secondary Outcome: WOMAC Total Score (Change From Baseline at Each Assessment Time Point)
Description: The WOMAC total subscale score was defined as the average of 24 items(5 pain subscale items, 17 physical functioning subscale items, and 2 stiffness subscale items). The participants assessed the past 48 hours on an 11-point numeric rating scale, from 0 (no stiffness) to 10(extremely stiffness), where smaller values being better.
Time Frame: Baseline to Week 68
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment Placebo | After the Amendment MT-5547 1 mg q8w | After the Amendment MT-5547 1 mg q4w
Number analyzed (Participants) | 204 | 203 | 165 | 162 | 165
units on a scale
  Week 1: number analyzed (Participants) | 203 | 203 | 165 | 162 | 165
  Week 1 | -0.46 (0.13) | -1.29 (0.13) | -0.42 (0.13) | -1.03 (0.14) | -1.18 (0.13)
  Week 2: number analyzed (Participants) | 201 | 200 | 162 | 162 | 162
  Week 2 | -0.60 (0.14) | -1.60 (0.14) | -0.56 (0.14) | -1.31 (0.14) | -1.47 (0.14)
  Week 4: number analyzed (Participants) | 201 | 201 | 163 | 162 | 163
  Week 4 | -0.78 (0.14) | -1.87 (0.15) | -0.75 (0.15) | -1.44 (0.15) | -1.70 (0.15)
  Week 8: number analyzed (Participants) | 199 | 200 | 161 | 160 | 162
  Week 8 | -1.02 (0.15) | -2.40 (0.15) | -0.98 (0.15) | -1.54 (0.16) | -2.23 (0.15)
  Week 12: number analyzed (Participants) | 193 | 197 | 155 | 158 | 159
  Week 12 | -1.31 (0.16) | -2.49 (0.16) | -1.28 (0.17) | -2.01 (0.17) | -2.31 (0.17)
  Week 16: number analyzed (Participants) | 190 | 189 | 152 | 158 | 152
  Week 16 | -1.46 (0.16) | -2.72 (0.16) | -1.45 (0.17) | -1.89 (0.17) | -2.56 (0.17)
  Week 20: number analyzed (Participants) | 189 | 185 | 151 | 157 | 150
  Week 20 | -2.10 (0.16) | -2.81 (0.16) | -2.03 (0.17) | -2.27 (0.17) | -2.60 (0.17)
  Week 24: number analyzed (Participants) | 186 | 180 | 148 | 149 | 146
  Week 24 | -2.28 (0.17) | -2.81 (0.17) | -2.24 (0.17) | -2.08 (0.17) | -2.68 (0.18)
  Week 28: number analyzed (Participants) | 184 | 177 | 146 | 143 | 143
  Week 28 | -2.23 (0.16) | -2.97 (0.17) | -2.20 (0.17) | -2.49 (0.17) | -2.83 (0.17)
  Week 32: number analyzed (Participants) | 180 | 175 | 142 | 142 | 141
  Week 32 | -2.30 (0.17) | -3.06 (0.17) | -2.31 (0.17) | -2.30 (0.17) | -2.89 (0.17)
  Week 36: number analyzed (Participants) | 173 | 173 | 135 | 136 | 139
  Week 36 | -2.37 (0.17) | -2.91 (0.17) | -2.39 (0.17) | -2.55 (0.17) | -2.75 (0.17)
  Week 40: number analyzed (Participants) | 170 | 171 | 133 | 133 | 137
  Week 40 | -2.36 (0.17) | -2.99 (0.17) | -2.36 (0.17) | -2.51 (0.18) | -2.80 (0.18)
  Week 44: number analyzed (Participants) | 170 | 162 | 133 | 134 | 129
  Week 44 | -2.42 (0.17) | -2.98 (0.17) | -2.44 (0.17) | -2.73 (0.17) | -2.78 (0.17)
  Week 48: number analyzed (Participants) | 170 | 161 | 133 | 132 | 128
  Week 48 | -2.45 (0.17) | -2.91 (0.18) | -2.42 (0.18) | -2.51 (0.18) | -2.70 (0.18)
  Week 52: number analyzed (Participants) | 167 | 160 | 131 | 133 | 127
  Week 52 | -2.08 (0.18) | -2.57 (0.18) | -2.11 (0.19) | -2.15 (0.19) | -2.33 (0.19)
  Week 60: number analyzed (Participants) | 163 | 156 | 127 | 131 | 123
  Week 60 | -2.24 (0.19) | -1.79 (0.19) | -2.29 (0.20) | -2.04 (0.20) | -1.57 (0.20)
  Week 68: number analyzed (Participants) | 162 | 151 | 126 | 130 | 121
  Week 68 | -2.20 (0.19) | -1.76 (0.19) | -2.29 (0.20) | -2.14 (0.20) | -1.57 (0.20)

7. Secondary Outcome: Patient Global Assessment (PGA) (Change From Baseline at Each Assessment Time Point)
Description: Patient Global Assessment(PGA) was a measure whereby the participant assessed global improvement in OA using the 5-level scale(1=very well; 2=well; 3=fair; 4=poor; and 5=very poor).
Time Frame: Baseline to Week 68
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled Placebo | Pooled MT-5547 1 mg q4w | After the Amendment Placebo | After the Amendment MT-5547 1 mg q8w | After the Amendment MT-5547 1 mg q4w
Number analyzed (Participants) | 204 | 203 | 165 | 162 | 165
units on a scale
  Week 1: number analyzed (Participants) | 203 | 203 | 165 | 162 | 165
  Week 1 | -0.3 (0.1) | -0.7 (0.1) | -0.4 (0.1) | -0.7 (0.1) | -0.7 (0.1)
  Week 2: number analyzed (Participants) | 201 | 200 | 162 | 162 | 162
  Week 2 | -0.5 (0.1) | -0.8 (0.1) | -0.5 (0.1) | -0.9 (0.1) | -0.8 (0.1)
  Week 4: number analyzed (Participants) | 201 | 201 | 163 | 162 | 163
  Week 4 | -0.5 (0.1) | -1.0 (0.1) | -0.5 (0.1) | -0.9 (0.1) | -1.0 (0.1)
  Week 8: number analyzed (Participants) | 199 | 200 | 161 | 160 | 162
  Week 8 | -0.6 (0.1) | -1.2 (0.1) | -0.7 (0.1) | -0.9 (0.1) | -1.2 (0.1)
  Week 12: number analyzed (Participants) | 194 | 197 | 156 | 158 | 159
  Week 12 | -0.8 (0.1) | -1.1 (0.1) | -0.8 (0.1) | -1.2 (0.1) | -1.1 (0.1)
  Week 16: number analyzed (Participants) | 190 | 189 | 152 | 158 | 152
  Week 16 | -0.8 (0.1) | -1.2 (0.1) | -0.9 (0.1) | -1.1 (0.1) | -1.2 (0.1)
  Week 20: number analyzed (Participants) | 189 | 185 | 151 | 157 | 150
  Week 20 | -1.1 (0.1) | -1.2 (0.1) | -1.1 (0.1) | -1.1 (0.1) | -1.2 (0.1)
  Week 24: number analyzed (Participants) | 186 | 180 | 148 | 149 | 146
  Week 24 | -1.2 (0.1) | -1.1 (0.1) | -1.2 (0.1) | -1.1 (0.1) | -1.2 (0.1)
  Week 28: number analyzed (Participants) | 184 | 177 | 146 | 143 | 143
  Week 28 | -1.0 (0.1) | -1.3 (0.1) | -1.1 (0.1) | -1.2 (0.1) | -1.3 (0.1)
  Week 32: number analyzed (Participants) | 180 | 175 | 142 | 142 | 141
  Week 32 | -1.1 (0.1) | -1.2 (0.1) | -1.1 (0.1) | -1.0 (0.1) | -1.2 (0.1)
  Week 36: number analyzed (Participants) | 173 | 173 | 135 | 136 | 139
  Week 36 | -1.2 (0.1) | -1.2 (0.1) | -1.2 (0.1) | -1.1 (0.1) | -1.2 (0.1)
  Week 40: number analyzed (Participants) | 170 | 171 | 133 | 133 | 137
  Week 40 | -1.1 (0.1) | -1.2 (0.1) | -1.1 (0.1) | -1.0 (0.1) | -1.2 (0.1)
  Week 44: number analyzed (Participants) | 170 | 162 | 133 | 134 | 129
  Week 44 | -1.2 (0.1) | -1.1 (0.1) | -1.2 (0.1) | -1.2 (0.1) | -1.1 (0.1)
  Week 48: number analyzed (Participants) | 170 | 161 | 133 | 132 | 128
  Week 48 | -1.1 (0.1) | -1.1 (0.1) | -1.1 (0.1) | -1.1 (0.1) | -1.1 (0.1)
  Week 52: number analyzed (Participants) | 167 | 160 | 131 | 133 | 127
  Week 52 | -0.9 (0.1) | -0.9 (0.1) | -0.9 (0.1) | -0.9 (0.1) | -0.9 (0.1)
  Week 60: number analyzed (Participants) | 163 | 156 | 127 | 131 | 123
  Week 60 | -0.9 (0.1) | -0.5 (0.1) | -1.0 (0.1) | -0.8 (0.1) | -0.5 (0.1)
  Week 68: number analyzed (Participants) | 162 | 151 | 126 | 130 | 121
  Week 68 | -0.9 (0.1) | -0.5 (0.1) | -1.0 (0.1) | -0.8 (0.1) | -0.6 (0.1)

8. Secondary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: Baseline to Week 68 (Treatment period=48 weeks, Post-treatment Observation Period=20weeks)
Population: The analysis was performed in the safety analysis set (SAF). The SAF consisted of all randomized participants except for the following participants
  * participants who did not receive study drug even once
  * participants for whom absolutely no post-randomization safety data are available
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo group is the same population as the Pooled Placebo group. Participants randomized to the Placebo group received MT-5547-matching placebo SC q4w from Week 0 to Week 44.
  Naproxen oral was received from the day after the Week 16 until Week 48.
- MT-5547 1 mg q8w: MT-5547 1mg q8w group is the same population as the After amendment MT-5547 1mg q8w.
  Participants randomized to the After the amendment MT-5547 1 mg q8w group received MT-5547 1 mg SC on Weeks 0, 8, 16, 24, 32, and 40, and MT-5547-matching placebo SC on Weeks 4, 12, 20, 28, 36, and 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 1mg q4w: MT-5547 1mg q4w group is the same population as the Pooled MT-5547 1mg q4w. Participants randomized to the Pooled MT-5547 1mg q4w group received MT-5547 1 mg SC q4w from Week 0 to Week 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 3 mg q4w: Participants randomized to the MT-5547 3 mg q4w group received MT-5547 3 mg SC q4w from Week 0 to Week 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 6 mg q8w: Participants randomized to the After the amendment MT-5547 6 mg q8w group received MT-5547 6 mg SC on Weeks 0, 8, 16, 24, 32, and 40, and MT-5547-matching placebo SC on Weeks 4, 12, 20, 28, 36, and 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
Arm/Group | Placebo | MT-5547 1 mg q8w | MT-5547 1mg q4w | MT-5547 3 mg q4w | MT-5547 6 mg q8w
Number analyzed (Participants) | 204 | 162 | 203 | 28 | 29
Participants
  Participants with at least one AE (Treatment Period) | 174 | 136 | 168 | 11 | 14
  Participants with at least one adverse drug reaction (treatment period) | 14 | 20 | 25 | 1 | 3
  Participants with at least one AE (post-treatment period) | 115 | 83 | 117 | 19 | 16
  Participants with at least one adverse drug reaction (post-treatment period) | 3 | 4 | 14 | 2 | 4

9. Secondary Outcome: Number of Participants With a Joint Replacement Procedure is Scheduled
Description: All the Joint Replacement surgeries that were performed within 20 weeks from the day after the end date of the treatment period were reported and tabulated in this study in order to assess the outcome of joint damage regardless of the presence or absence of related adjudicated arthropathy. The subjects who were going to undergo JR surgery were to be withdrawn from study treatment.
Time Frame: Baseline to Week 68
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT-5547 1 mg q8w | MT-5547 1mg q4w | MT-5547 3 mg q4w | MT-5547 6 mg q8w
Number analyzed (Participants) | 204 | 162 | 203 | 28 | 29
Participants | 4 | 5 | 10 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 68 (Treatment period=48 weeks, Post-treatment Observation Period=20weeks)
Description: The analysis of safety was performed in the safety analysis set (SAF). The SAF consisted of all randomized participants except for the following participants
  * participants who did not receive study drug even once
  * participants for whom absolutely no post-randomization safety data are available Reported AEs & deaths are treatment emergent.
Groups:
- Placebo, On-treatment Period; Placebo, Post-treatment Observation Period: Placebo group is the same population as the Pooled Placebo group. Participants randomized to the Placebo group received MT-5547-matching placebo SC q4w from Week 0 to Week 44.
  Naproxen oral was received from the day after the Week 16 until Week 48.
- MT-5547 1 mg q8w, On-treatment Period; MT-5547 1 mg q8w, Post-treatment Observation Period: MT-5547 1mg q8w group is the same population as the After amendment MT-5547 1mg q8w.
  Participants randomized to the After the amendment MT-5547 1 mg q8w group received MT-5547 1 mg SC on Weeks 0, 8, 16, 24, 32, and 40, and MT-5547-matching placebo SC on Weeks 4, 12, 20, 28, 36, and 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 1mg q4w, On-treatment Period; MMT-5547 1mg q4w, Post-treatment Observation Period: MT-5547 1mg q4w group is the same population as the Pooled MT-5547 1mg q4w. Participants randomized to the Pooled MT-5547 1mg q4w group received MT-5547 1 mg SC q4w from Week 0 to Week 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 3 mg q4w, On-treatment Period; MT-5547 3 mg q4w, Post-treatment Observation Period: Participants randomized to the MT-5547 3 mg q4w group received MT-5547 3 mg SC q4w from Week 0 to Week 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
- MT-5547 6 mg q8w, On-treatment Period; MT-5547 6 mg q8w, Post-treatment Observation Period: Participants randomized to the After the amendment MT-5547 6 mg q8w group received MT-5547 6 mg SC on Weeks 0, 8, 16, 24, 32, and 40, and MT-5547-matching placebo SC on Weeks 4, 12, 20, 28, 36, and 44.
  Naproxen-matching placebo oral was received from the day after the Week 16 until Week 48.
Arm/Group | Placebo, On-treatment Period | MT-5547 1 mg q8w, On-treatment Period | MT-5547 1mg q4w, On-treatment Period | MT-5547 3 mg q4w, On-treatment Period | MT-5547 6 mg q8w, On-treatment Period | Placebo, Post-treatment Observation Period | MT-5547 1 mg q8w, Post-treatment Observation Period | MMT-5547 1mg q4w, Post-treatment Observation Period | MT-5547 3 mg q4w, Post-treatment Observation Period | MT-5547 6 mg q8w, Post-treatment Observation Period
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/162 | 0/203 | 0/28 | 0/29 | 0/204 | 0/162 | 0/203 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 6/204 | 4/162 | 9/203 | 0/28 | 0/29 | 5/204 | 3/162 | 7/203 | 3/28 | 3/29
Other Adverse Events (participants affected / at risk) | 108/204 | 85/162 | 118/203 | 4/28 | 11/29 | 51/204 | 37/162 | 65/203 | 12/28 | 7/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo, On-treatment Period (N=204) | MT-5547 1 mg q8w, On-treatment Period (N=162) | MT-5547 1mg q4w, On-treatment Period (N=203) | MT-5547 3 mg q4w, On-treatment Period (N=28) | MT-5547 6 mg q8w, On-treatment Period (N=29) | Placebo, Post-treatment Observation Period (N=204) | MT-5547 1 mg q8w, Post-treatment Observation Period (N=162) | MMT-5547 1mg q4w, Post-treatment Observation Period (N=203) | MT-5547 3 mg q4w, Post-treatment Observation Period (N=28) | MT-5547 6 mg q8w, Post-treatment Observation Period (N=29)
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corticobasal degeneration (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo, On-treatment Period (N=204) | MT-5547 1 mg q8w, On-treatment Period (N=162) | MT-5547 1mg q4w, On-treatment Period (N=203) | MT-5547 3 mg q4w, On-treatment Period (N=28) | MT-5547 6 mg q8w, On-treatment Period (N=29) | Placebo, Post-treatment Observation Period (N=204) | MT-5547 1 mg q8w, Post-treatment Observation Period (N=162) | MMT-5547 1mg q4w, Post-treatment Observation Period (N=203) | MT-5547 3 mg q4w, Post-treatment Observation Period (N=28) | MT-5547 6 mg q8w, Post-treatment Observation Period (N=29)
Cataract (Eye disorders) | 3 | 0 | 4 | 0 | 0 | 2 | 0 | 1 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 6 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 59 | 49 | 62 | 2 | 4 | 25 | 12 | 14 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 17 | 9 | 12 | 0 | 2 | 2 | 5 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8 | 17 | 0 | 0 | 8 | 2 | 7 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 14 | 17 | 0 | 0 | 7 | 2 | 4 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3 | 2 | 0 | 1 | 1 | 5 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 0 | 10 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 5 | 3 | 5 | 0 | 0 | 5 | 7 | 11 | 0 | 0
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 7 | 20 | 0 | 1 | 1 | 4 | 17 | 2 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 4 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 3 | 8 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 23 | 15 | 16 | 0 | 0 | 2 | 2 | 4 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT03245008/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT03245008/SAP_001.pdf